CLINICAL TRIAL: NCT05098093
Title: Bioavailabity of the Major Metabolites of a Botanical Extract, in Healthy Adults : a Randomized, Cross-over, Open-label, Clinical Study
Brief Title: Bioavailabity of the Major Metabolites of a Botanical Extract, in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Collaborators: CIC Inserm 1405, University Hospital Clermont-Ferrand, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIODAI-2021
Record Dates: First submitted 2021-10-06; First posted 2021-10-28 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized botanical extract (Active Comparator)
  Interventions: Dietary Supplement: SBE
- Dry botanical extract (Active Comparator)
  Interventions: Dietary Supplement: DBE
- Botanical powder (Active Comparator)
  Interventions: Dietary Supplement: BP

INTERVENTIONS:
Dietary Supplement: SBE — Hard-shell capsule
  Arms: Standardized botanical extract
Dietary Supplement: DBE — Hard-shell capsule
  Arms: Dry botanical extract
Dietary Supplement: BP — Hard-shell capsule
  Arms: Botanical powder

SUMMARY:
Scientific research on the beneficial effects of botanical extracts has led to a better understanding of the role of its bioactive compounds, but the bioavailability in human remains largely unknown. Indeed, the most of publications investigated the bioavailability of metabolites of spices in in vitro cells model or animal experiments but few clinical studies have been conducted.

Therefore, the aim of this study is to characterize and quantify in blood, the main metabolite compounds of a botanical extract, following its administration by different routes (oral or sublingual) and with different preparations (extract or powder), in quantity equivalent to those having demonstrated biological properties.

ELIGIBILITY:
Inclusion Criteria:

* Male adults
* Age between 18 and 35 years (limits included);
* Non-smoking individuals (nor tobacco, nor electronic cigarette nor cannabis, former smokers can be included if they stopped smoking at least 2 years ago);
* Body Mass Index ≥ 19 and < 30 kg/m2.
* Considered healthy based on their medical history, clinical examination and biological examination;
* Subjects capable of and willing to comply with the protocol and to give their written informed consent.
* Subjects affiliated with a social security scheme.

Non-inclusion Criteria:

Subjects complying with at least one of the following criteria will not be eligible:

* Known metabolic abnormality or clinically significant medical condition, such as:

  * Cardiovascular disease (other than hypertension),
  * Neurological disease,
  * Psychatric disease,
  * Immunological disease,
  * Endocrine disease (including diabetes or thyroid diseases),
  * Chronic kidney disease,
  * Heamatological abnormalities
* Hypertension (SBP≥160 mm Hg or DBP ≥100 mm Hg).
* Use of any type of medication or narcotic drug (detected either by the self-declaration of the participant and/ or by the urine TetraHydroCannabinol (THC) test) currently or within the past 2 months before entry into the study;
* Self-reported alcohol intake of >10 units/ week
* Weight changes above 10% body weight within the past 6 months before entering the study;
* Currently under prescribed diet regimen, whatever the reason;
* Consumption of food supplement(s) currently or within the past 4 weeks before entry into the study, such as but not limited to: botanicals, vitamins, minerals, amino acids; anti-oxydant;
* Any intolerance or allergy documented or suspected to one of the components of the study products;
* Subject presenting a psychological or linguistic inability to sign the informed consent;
* Subject under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Subject participating in another biomedical study or participation in another study where a product (ie: dietary supplement) were consumed within the 3 months before entry into this study;
* Any regulatory reason according to national applicable regulation;
* Subject having received indemnities for clinical trial reaching at least 4500 Euros considering the last 12 months.

Exclusion criteria :

During the study, in case of emergence of a new health condition or treatment considered as non-inclusion criteria or likely to affect the study parameters according to Investigator's judgment, the participants will be excluded from the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
(AUC 0-t) : Area under the curve of the serum concentration of the main metabolites of the products. | From 0 to 180 min after product ingestion

SECONDARY OUTCOMES:
AUC 0-t for the main metabolites of the products. | From 0 to 180 min after product ingestion
  Comparison between tested products
Serum peak concentration (Cmax) of the metabolites of the tested products. | From 0 to 180 min after product ingestion
  Determination and comparison between products
Time to serum peak concentration (Tmax) of the metabolites of the tested products. | From 0 to 180 min after product ingestion
  Determination and comparison between products
Elimination half-life (T1/2) of serum metabolites of the tested products defined by the time required for the concentration of product metabolites to decrease to half of Cmax. | From 0 to 180 min after product ingestion
  Determination and comparison between products
Concentration of urinary crocetin (ng/mg of creatinine) of the tested products at the end of the visit | 185 min after product intake
  Determination and comparison between products
Systolic and diastolic blood pressure | 183 min after product ingestion
  Comparison between tested products

OTHER OUTCOMES:
AUC(0-t) of the main volatile metabolite of the tested products in serum | From 0 to 180 min after product ingestion
  Determination and comparison between SBE and DBE
Cmax of the main volatile metabolite of the tested products in serum | From 0 to 180 min after product ingestion
  Determination and comparison between SBE and DBE
Tmax of the main volatile metabolite of the tested products in serum | From 0 to 180 min after product ingestion
  Determination and comparison between SBE and DBE
T1/2 of the main volatile metabolite of the tested products in serum | From 0 to 180 min after product ingestion
  Determination and comparison between SBE and DBE

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Inserm 1405, University Hospital Clermont-Ferrand,, Clermont-Ferrand, France